CLINICAL TRIAL: NCT02963506
Title: A Multicenter, Phase 2B, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study to Evaluate the Efficacy and Safety of Bimekizumab in Subjects With Active Ankylosing Spondylitis
Brief Title: A Study to Evaluate the Efficacy and Safety of Different Doses of Bimekizumab in Subjects With Active Ankylosing Spondylitis
Acronym: BE AGILE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS0008; 2016-001102-42 (EudraCT Number)
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Ankylosing Spondylitis
Keywords: AS; Ankylosing Spondylitis; Bimekizumab
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Subjects will receive for 12 Weeks Placebo and will then be re-randomized to Bimekizumab Dose 3 or Bimekizumab Dose 4 for 36 Weeks.
  Interventions: Other: Placebo
- Bimekizumab Dose 1 (Experimental): Subjects will receive for 12 Weeks Bimekizumab Dose 1 and will then be re-randomized to Bimekizumab Dose 3 or Bimekizumab Dose 4 for 36 Weeks.
  Interventions: Drug: Bimekizumab
- Bimekizumab Dose 2 (Experimental): Subjects will receive for 12 Weeks Bimekizumab Dose 2 and will then be re-randomized to Bimekizumab Dose 3 or Bimekizumab Dose 4 for 36 Weeks.
  Interventions: Drug: Bimekizumab
- Bimekizumab Dose 3 (Experimental): Subjects will receive for 48 Weeks Bimekizumab Dose 3.
  Interventions: Drug: Bimekizumab
- Bimekizumab Dose 4 (Experimental): Subjects will receive for 48 Weeks Bimekizumab Dose 4.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Other: Placebo
  Arms: Placebo
Drug: Bimekizumab — Bimekizumab in different dosages.
  Other Names: UCB4940
  Arms: Bimekizumab Dose 1; Bimekizumab Dose 2; Bimekizumab Dose 3; Bimekizumab Dose 4

SUMMARY:
This is a study to evaluate the efficacy and safety of different doses of bimekizumab in subjects with active Ankylosing Spondylitis (AS).

ELIGIBILITY:
Inclusion Criteria:

* Subject has active ankylosing spondylitis (AS), determined by documented radiologic evidence fulfilling the Modified New York criteria for AS including symptoms for >=3 months and age of onset <45 years
* Subject has moderate to severe active disease as defined by each of the following:

  1. BASDAI score >=4
  2. Spinal pain >=4 on a 0 to 10 NRS (Numeric Rating Scale; from BASDAI item 2)
* Subjects must have at least 1 of the following:

  1. inadequate response to nonsteroidal anti-inflammatory drug (NSAID) therapy
  2. intolerance to administration of at least 1 NSAID
  3. contraindication(s) to NSAID therapy
* Subjects who are regularly taking NSAIDs/COX-2 inhibitors as part of their AS therapy are required to be on a stable dose for at least 14 days before Baseline
* Subjects taking corticosteroids must be on an average daily dose of <=10mg/day prednisone or equivalent for at least 14 days before Baseline and should remain on a stable dose up to Week 16
* Subjects taking methotrexate (MTX) (<=25mg/week) are allowed to continue their medication if started at least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomization
* Subjects taking sulfasalazine (up to 3grams/day) or hydroxychloroquine (up to 400mg per day total) are allowed to continue their medication if started at least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomization
* Subjects may be tumor necrosis factor (TNF) inhibitor-naïve or may have received 1 prior TNF inhibitor. Subjects who have been on a TNF inhibitor previously must have:

  1. experienced an inadequate response to previous treatment given for at least 12 weeks
  2. been intolerant to administration (eg, had a side effect/adverse event that led to discontinuation)
  3. lost access to TNF inhibitor for other reasons

Exclusion Criteria:

* Subjects with a total ankylosis of the spine, or a diagnosis of any other inflammatory arthritis eg, rheumatoid arthritis (RA), sarcoidosis, systemic lupus erythematosus, or reactive arthritis
* Subjects with any current sign or symptom that may indicate an active infection (except for the common cold)
* Subjects with a history of chronic or recurrent infections, or a serious or life-threatening infection within the 6 months prior to the Baseline Visit
* Subjects receiving any live vaccination within the 8 weeks prior to Baseline
* Subjects with known tuberculosis (TB) infection, at high risk of acquiring TB infection, with latent TB infection or current or history of nontuberculous mycobacteria (NTMB) infection
* Subjects with concurrent malignancy or a history of malignancy during the past 5 years will be excluded, with following exceptions that may be included:

  1. <= 3 excised or ablated basal cell carcinomas of the skin
  2. One squamous cell carcinoma of the skin (stage T1 maximum) successfully excised, or ablated only (other treatments, ie, chemotherapy, do not apply), with no signs of recurrence or metastases for more than 2 years prior to Screening
  3. Actinic keratosis (-es)
  4. Squamous cell carcinoma-in-situ of the skin successfully excised, or ablated, more than 6 months prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273(UCB)
Locations (74):
- United States (15):
  - As0008 019, Anniston, Alabama
  - As0008 007, La Jolla, California
  - As0008 009, Upland, California
  - As0008 005, Aventura, Florida
  - As0008 022, Ormond Beach, Florida
  - As0008 030, Sarasota, Florida
  - As0008 027, Boston, Massachusetts
  - As0008 021, Freehold, New Jersey
  - As0008 015, Cleveland, Ohio
  - As0008 014, Portland, Oregon
  - As0008 001, Duncansville, Pennsylvania
  - As0008 020, Austin, Texas
  - As0008 006, Dallas, Texas
  - As0008 018, Houston, Texas
  - As0008 002, Seattle, Washington
- Bulgaria (5):
  - As0008 156, Dobrich
  - As0008 151, Plovdiv
  - As0008 154, Plovdiv
  - As0008 155, Plovdiv
  - As0008 150, Rousse
- Canada (3):
  - As0008 101, Québec
  - As0008 100, Victoria
  - As0008 103, Winnipeg
- Czechia (10):
  - As0008 205, Brno
  - As0008 206, Hustopeče
  - As0008 207, Olomouc
  - As0008 208, Pardubice
  - As0008 201, Prague
  - As0008 202, Prague
  - As0008 209, Prague
  - As0008 210, Prague
  - As0008 211, Prague
  - As0008 203, Zlín
- Germany (5):
  - As0008 302, Cologne
  - As0008 304, Hamburg
  - As0008 308, Hanover
  - As0008 303, Herne
  - As0008 301, Ratingen
- Hungary (4):
  - As0008 400, Budapest
  - As0008 403, Budapest
  - As0008 402, Debrecen
  - As0008 401, Veszprém
- Poland (14):
  - As0008 466, Bydgoszcz
  - As0008 453, Elblag
  - As0008 456, Elblag
  - As0008 455, Krakow
  - As0008 461, Lublin
  - As0008 467, Nowa Sól
  - As0008 451, Poznan
  - As0008 462, Poznan
  - As0008 450, Torun
  - As0008 454, Warsaw
  - As0008 459, Warsaw
  - As0008 457, Wroclaw
  - As0008 460, Wroclaw
  - As0008 465, Wroclaw
- Russia (9):
  - As0008 601, Moscow
  - As0008 604, Moscow
  - As0008 605, Moscow
  - As0008 607, Moscow
  - As0008 600, Saint Petersburg
  - As0008 606, Saint Petersburg
  - As0008 608, Saint Petersburg
  - As0008 609, Saint Petersburg
  - As0008 610, Saint Petersburg
- Spain (3):
  - As0008 801, A Coruña
  - As0008 800, Córdoba
  - As0008 803, Santiago de Compostela
- Ukraine (6):
  - As0008 700, Kiev
  - As0008 707, Kyiv
  - As0008 705, Ternopil
  - As0008 708, Uzhhorod
  - As0008 706, Vinnytsia
  - As0008 704, Zaporizhya

REFERENCES:
- [Result] van der Heijde D, Gensler LS, Deodhar A, Baraliakos X, Poddubnyy D, Kivitz A, Farmer MK, Baeten D, Goldammer N, Coarse J, Oortgiesen M, Dougados M. Dual neutralisation of interleukin-17A and interleukin-17F with bimekizumab in patients with active ankylosing spondylitis: results from a 48-week phase IIb, randomised, double-blind, placebo-controlled, dose-ranging study. Ann Rheum Dis. 2020 May;79(5):595-604. doi: 10.1136/annrheumdis-2020-216980. Epub 2020 Apr 6. PMID 32253184
- [Result] Robinson PC, Machado PM, Haroon N, Gensler LS, Reveille JD, Taieb V, Vaux T, Fleurinck C, Oortgiesen M, de Peyrecave N, Deodhar A. Minimal Impact of the COVID-19 Pandemic on Disease Activity and Health-Related Quality of Life in Patients With Ankylosing Spondylitis Receiving Bimekizumab: Exploratory Analyses From a Phase 2b Open-Label Extension Study. ACR Open Rheumatol. 2022 Sep;4(9):819-824. doi: 10.1002/acr2.11486. Epub 2022 Jul 14. PMID 35833532
- [Derived] Mease PJ, Gensler LS, Orbai AM, Warren RB, Bajracharya R, Ink B, Marten A, Massow U, Shende V, Manente M, Peterson L, White K, Landewe R, Poddubnyy D. Long-term safety of bimekizumab in adult patients with axial spondyloarthritis or psoriatic arthritis: pooled results from integrated phase IIb/III clinical studies. RMD Open. 2025 Apr 6;11(2):e005026. doi: 10.1136/rmdopen-2024-005026. PMID 40194794
- [Derived] Deodhar A, Navarro-Compan V, Poddubnyy D, Gensler LS, Ramiro S, Tomita T, Marzo-Ortega H, Fleurinck C, Vaux T, Massow U, de Peyrecave N, van der Heijde D, Baraliakos X. Long-term safety and sustained efficacy of bimekizumab in patients with ankylosing spondylitis (radiographic axial spondyloarthritis): 5-year results from BE AGILE (phase 2b) and its open-label extension. RMD Open. 2025 Jan 31;11(1):e005081. doi: 10.1136/rmdopen-2024-005081. PMID 39890205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in October 2016 and concluded in August 2018.
Pre-assignment Details: The study included a 28-Day Screening Period, followed by a Double-Blind Period from Day 1 to Week 12, prior to treatment re-randomization, a Dose-blind Period, from Week 12 after the treatment re-randomization and up to Week 48 and a Safety Follow-Up (SFU) Period, post Week 48.
  The Participant Flow refers to the Randomized Set and Dose-Blind Set.
Groups:
- Placebo: Participants received placebo during the 12 weeks Double-Blind Period.
- BKZ 16 mg: Participants received bimekizumab (BKZ) 16 milligrams (mg) every 4 weeks (Q4W) during the 12 weeks Double-Blind Period.
- BKZ 64 mg: Participants received bimekizumab (BKZ) 64 mg every 4 weeks (Q4W) during the 12 weeks Double-Blind Period.
- BKZ 160 mg: Participants received bimekizumab (BKZ) 160 mg every 4 weeks (Q4W) during the 12 weeks Double-Blind Period followed by the same dose during the 36 weeks Dose-Blind Period.
- BKZ 320 mg: Participants received bimekizumab (BKZ) 320 mg every 4 weeks (Q4W) during the 12 weeks Double-Blind Period followed by the same dose during the 36 weeks Dose-Blind Period.
- Placebo - BKZ 160 mg: After the 12 weeks Double-Blind Period participants randomized to placebo were re-randomized to receive bimekizumab (BKZ) 160 mg every 4 weeks (Q4W) for 36 weeks in the Dose-Blind Period.
- Placebo - BKZ 320 mg: After the 12 weeks Double-Blind Period participants randomized to placebo were re-randomized to receive bimekizumab (BKZ) 320 mg every 4 weeks (Q4W) for 36 weeks in the Dose-Blind Period
- BKZ 16 mg - BKZ 160 mg: After the 12 weeks Double-Blind Period participants randomized to bimekizumab (BKZ) 16 mg every 4 weeks (Q4W) were re-randomized to receive BKZ 160 mg Q4W for 36 weeks in the Dose-Blind Period.
- BKZ 16 mg - BKZ 320 mg: After the 12 weeks Double-Blind Period participants randomized to bimekizumab (BKZ) 16 mg every 4 weeks (Q4W) were re-randomized to receive BKZ 320 mg Q4W for 36 weeks in the Dose-Blind Period.
- BKZ 64 mg - BKZ 160 mg: After the 12 weeks Double-Blind Period participants randomized to bimekizumab (BKZ) 64 mg every 4 weeks (Q4W) were re-randomized to receive BKZ 160 mg Q4W for 36 weeks in the Dose-Blind Period.
- BKZ 64 mg - BKZ 320 mg: After the 12 weeks Double-Blind Period participants randomized to bimekizumab (BKZ) 64 mg every 4 weeks (Q4W) were re-randomized to receive BKZ 320 mg Q4W for 36 weeks in the Dose-Blind Period.
- BKZ 160 mg - BKZ 160 mg: Participants randomized to bimekizumab (BKZ) 160 mg every 4 weeks (Q4W) in the 12 weeks Double-Blind Period, continued to receive BKZ 160 mg Q4W in the 36 weeks Dose-Blind Period.
- BKZ 320 mg - BKZ 320 mg: Participants randomized to bimekizumab (BKZ) 320 mg every 4 weeks (Q4W) in the 12 weeks Double-Blind Period, continued to receive BKZ 320 mg Q4W in the 36 weeks Dose-Blind Period.
Period: Double-Blind Period
Arm/Group | Placebo | BKZ 16 mg | BKZ 64 mg | BKZ 160 mg | BKZ 320 mg | Placebo - BKZ 160 mg | Placebo - BKZ 320 mg | BKZ 16 mg - BKZ 160 mg | BKZ 16 mg - BKZ 320 mg | BKZ 64 mg - BKZ 160 mg | BKZ 64 mg - BKZ 320 mg | BKZ 160 mg - BKZ 160 mg | BKZ 320 mg - BKZ 320 mg
Started | 60 | 61 | 61 | 60 | 61 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Double-Blind Period | 60 | 59 | 59 | 58 | 61 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Week 12 - Started Dose-Blind | 60 | 58 | 59 | 58 | 61 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 60 | 58 | 59 | 58 | 61 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No compliance | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse event, non fatal after Wk12 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose-Blind Period
Arm/Group | Placebo | BKZ 16 mg | BKZ 64 mg | BKZ 160 mg | BKZ 320 mg | Placebo - BKZ 160 mg | Placebo - BKZ 320 mg | BKZ 16 mg - BKZ 160 mg | BKZ 16 mg - BKZ 320 mg | BKZ 64 mg - BKZ 160 mg | BKZ 64 mg - BKZ 320 mg | BKZ 160 mg - BKZ 160 mg | BKZ 320 mg - BKZ 320 mg
Started | 0 | 0 | 0 | 0 | 0 | 24 | 36 | 31 | 27 | 34 | 25 | 58 | 61
Completed | 0 | 0 | 0 | 0 | 0 | 20 | 31 | 26 | 24 | 30 | 24 | 56 | 54
Not Completed | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 5 | 3 | 4 | 1 | 2 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 2 | 2 | 1 | 1 | 6
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Sponsor decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Meeting exclusion criteria 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refer to the Full Analysis Set (FAS), which consisted all randomized study participants who received at least 1 dose of investigational medicinal product (IMP) and had a valid measurement of the primary efficacy variable at Baseline.
Arm/Group | Placebo | BKZ 16 mg | BKZ 64 mg | BKZ 160 mg | BKZ 320 mg | Total Title
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 61 | 303
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 56 | 59 | 56 | 60 | 291
  >=65 years | 0 | 5 | 2 | 4 | 1 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.65 (10.30) | 43.31 (12.59) | 40.41 (10.93) | 42.38 (13.11) | 45.02 (11.39) | 42.16 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 9 | 8 | 11 | 47
  Male | 49 | 53 | 52 | 52 | 50 | 256
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 0 | 0 | 1 | 0 | 0 | 1
  White | 60 | 58 | 60 | 59 | 61 | 298
  Other/Mixed | 0 | 3 | 0 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Axial Spondyloarthritis International Society 40% Response Criteria (ASAS40) at Week 12
Description: The ASAS40 response was defined as relative improvements of at least 40% and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS), where 0 is "not active" and 10 is "very active" in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS score), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain.
  Note: Participants with missing data or who discontinue study treatment prior to Week 12 were counted as non-responders.
Time Frame: Week 12
Population: The FAS consisted of all randomized participants who received at least 1 dose of investigational medicinal product (IMP) and had a valid measurement of the primary efficacy variable at Baseline.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (FAS): Participants received placebo during the 12 weeks Double-Blind Period, forming the Full Analysis Set (FAS).
- BKZ 16 mg (FAS): Participants received bimekizumab (BKZ) 16 milligrams (mg) every 4 weeks (Q4W) during the 12 weeks Double-Blind Period, forming the Full Analysis Set (FAS).
- BKZ 64 mg (FAS): Participants received bimekizumab (BKZ) 64 mg every 4 weeks (Q4W) during the 12 weeks Double-Blind Period, forming the Full Analysis Set (FAS).
- BKZ 160 mg (FAS): Participants received bimekizumab (BKZ) 160 mg every 4 weeks (Q4W) during the 12 weeks Double-Blind Period followed by the same dose during the 36 weeks Dose-Blind Period, forming the Full Analysis Set (FAS).
- BKZ 320 mg (FAS): Participants received bimekizumab (BKZ) 320 mg every 4 weeks (Q4W) during the 12 weeks Double-Blind Period followed by the same dose during the 36 weeks Dose-Blind Period, forming the Full Analysis Set (FAS).
Arm/Group | Placebo (FAS) | BKZ 16 mg (FAS) | BKZ 64 mg (FAS) | BKZ 160 mg (FAS) | BKZ 320 mg (FAS)
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 61
percentage of participants | 13.3 | 29.5 | 42.6 | 46.7 | 45.9
Statistical Analysis 1: Comparison: Placebo (FAS) vs BKZ 16 mg (FAS) vs BKZ 64 mg (FAS) vs BKZ 160 mg (FAS) vs BKZ 320 mg (FAS); Statistic and p-value were calculated using a Cochran-Mantel-Haenszel test (test for non-zero correlation statistic) based on modified ridit scores and including geographic region and prior Tumor Necrosis Factor (TNF) inhibitor exposure as stratification factors; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Correlation statistic = 17.9
Statistical Analysis 2: Comparison: Placebo (FAS) vs BKZ 16 mg (FAS); For differences in relation to placebo: Odds Ratio, confidence interval and p-value were derived from a logistic regression model including fixed effects for treatment, geographic region and prior tumor necrosis factor (TNF) inhibitor exposure; Test type: Other — The pairwise testing of each bimekizumab dose versus placebo accounted for multiplicity by using a fixed sequence testing procedure with each bimekizumab dose being tested sequentially from the highest dose to the lowest dose. If the sequential testing failed to reach significance at a significance level of alpha=0.05, then the pairwise testing continued and the comparison was seen as non-significant; p = 0.040, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 2.6, 95% CI 2-sided [1.04 to 6.48]
Statistical Analysis 3: Comparison: Placebo (FAS) vs BKZ 64 mg (FAS); For differences in relation to placebo: Odds Ratio, confidence interval and p-value were derived from a logistic regression model including fixed effects for treatment, geographic region and prior TNF inhibitor exposure; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.001, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 4.5, 95% CI 2-sided [1.83 to 10.86]
Statistical Analysis 4: Comparison: Placebo (FAS) vs BKZ 160 mg (FAS); [analysis description as in outcome 1, analysis 3]; Test type: Other — [test comment as in outcome 1, analysis 2]; p < 0.001, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 5.5, 95% CI 2-sided [2.27 to 13.48]
Statistical Analysis 5: Comparison: Placebo (FAS) vs BKZ 320 mg (FAS); [analysis description as in outcome 1, analysis 3]; Test type: Other — [test comment as in outcome 1, analysis 2]; p < 0.001, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 5.3, 95% CI 2-sided [2.19 to 12.92]

2. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score - C-Reactive Protein (ASDAS [CRP]) at Week 12
Description: The ASDAS was calculated as the sum of the following components:
  0.121 x Back pain (BASDAI question 2 result) 0.058 x Duration of morning stiffness (BASDAI question 6 result) 0.110 x PGADA 0.073 x Peripheral pain/swelling (BASDAI question 3 result) 0.579 x (natural logarithm of the (hs-CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue are all assessed on a numerical scale (0 to 10 units).
  The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening. There is a minimum score of 0.636 for the total ASDAS score, but no defined upper score since CRP does not have a set upper limit.
  If one component for the ASDAS-CRP was missing at a given visit, that component was imputed by carrying the last observation forward, and the ASDAS-CRP was calculated accordingly. If the hs-CRP value was below 2 mg/L, then it was imputed as the constant value of 2 mg/L.
Time Frame: From Baseline to Week 12
Population: The FAS consisted of all randomized participants who received at least 1 dose of IMP and had a valid measurement of the primary efficacy variable at Baseline.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (FAS) | BKZ 16 mg (FAS) | BKZ 64 mg (FAS) | BKZ 160 mg (FAS) | BKZ 320 mg (FAS)
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 61
scores on a scale | -0.3 (0.17) | -0.8 (0.17) | -1.4 (0.17) | -1.3 (0.17) | -1.4 (0.17)
Statistical Analysis 1: Comparison: Placebo (FAS) vs BKZ 16 mg (FAS); Least squares (LS) Mean, standard error, confidence interval and p-value were derived using the analysis of covariance (ANCOVA) model with treatment, geographic region and prior TNF inhibitor exposure as fixed effects and the Baseline value as covariate; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference vs placebo = -0.5, 95% CI 2-sided [-0.86 to -0.24], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Placebo (FAS) vs BKZ 64 mg (FAS); LS Mean, standard error, confidence interval and p-value were derived using the ANCOVA model with treatment, geographic region and prior TNF inhibitor exposure as fixed effects and the Baseline value as covariate; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference vs placebo = -1.2, 95% CI 2-sided [-1.47 to -0.83], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Placebo (FAS) vs BKZ 160 mg (FAS); [analysis description as in outcome 2, analysis 2]; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference vs placebo = -1.0, 95% CI 2-sided [-1.35 to -0.72], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Placebo (FAS) vs BKZ 320 mg (FAS); [analysis description as in outcome 2, analysis 2]; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference vs placebo = -1.1, 95% CI 2-sided [-1.45 to -0.82], Standard Error of Mean 0.16

3. Secondary Outcome: Percentage of Participants With Axial Spondyloarthritis International Society 20% Response Criteria (ASAS20) at Week 12
Description: The ASAS20 response was defined as an improvement of at least 20% and absolute improvement of at least 1 unit on a 0 to 10 NRS, where 0 is "not active" and 10 is "very active" in at least 3 of the 4 domains: PGADA, Pain assessment (total spinal pain NRS scores), Function (BASFI), Inflammation (mean of BASDAI questions 5 and 6 concerning morning stiffness intensity and duration) and absence of deterioration in the potential remaining domain [deterioration was defined as a relative worsening of at least 20% and an absolute worsening of at least 1 unit].
  Note: Participants with missing data or who discontinue study treatment prior to Week 12 were counted as non-responders.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | BKZ 16 mg (FAS) | BKZ 64 mg (FAS) | BKZ 160 mg (FAS) | BKZ 320 mg (FAS)
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 61
percentage of participants | 28.3 | 41.0 | 62.3 | 58.3 | 72.1
Statistical Analysis 1: Comparison: Placebo (FAS) vs BKZ 16 mg (FAS); [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.163, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.80 to 3.67]
Statistical Analysis 2: Comparison: Placebo (FAS) vs BKZ 64 mg (FAS); [analysis description as in outcome 1, analysis 3]; Test type: Other; p < 0.001, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 3.9, 95% CI 2-sided [1.84 to 8.48]
Statistical Analysis 3: Comparison: Placebo (FAS) vs BKZ 160 mg (FAS); [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.001, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 3.5, 95% CI 2-sided [1.66 to 7.61]
Statistical Analysis 4: Comparison: Placebo (FAS) vs BKZ 320 mg (FAS); [analysis description as in outcome 1, analysis 3]; Test type: Other; p < 0.001, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 6.5, 95% CI 2-sided [2.92 to 14.28]

4. Secondary Outcome: Percentage of Participants With Axial Spondyloarthritis International Society (ASAS) 5/6 Response at Week 12
Description: The ASAS 5/6 response was defined as at least 20% improvement in at least 5 of the 6 domains: PGADA, Pain assessment (total spinal pain NRS scores), Function (BASFI), Inflammation (mean of BASDAI questions 5 and 6 concerning morning stiffness intensity and duration), spinal mobility (lateral spinal flexion) and high sensitivity C-reactive protein (hs-CRP).
  Note: Participants with missing data or who discontinue study treatment prior to Week 12 were counted as non-responders.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | BKZ 16 mg (FAS) | BKZ 64 mg (FAS) | BKZ 160 mg (FAS) | BKZ 320 mg (FAS)
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 61
percentage of participants | 6.7 | 29.5 | 49.2 | 53.3 | 54.1
Statistical Analysis 1: Comparison: Placebo (FAS) vs BKZ 16 mg (FAS); [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.003, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 5.3, 95% CI 2-sided [1.74 to 15.96]
Statistical Analysis 2: Comparison: Placebo (FAS) vs BKZ 64 mg (FAS); [analysis description as in outcome 1, analysis 3]; Test type: Other; p < 0.001, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 11.9, 95% CI 2-sided [4.03 to 35.38]
Statistical Analysis 3: Comparison: Placebo (FAS) vs BKZ 160 mg (FAS); [analysis description as in outcome 1, analysis 3]; Test type: Other; p < 0.001, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 14.3, 95% CI 2-sided [4.81 to 42.46]
Statistical Analysis 4: Comparison: Placebo (FAS) vs BKZ 320 mg (FAS); [analysis description as in outcome 1, analysis 3]; Test type: Other; p < 0.001, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 14.9, 95% CI 2-sided [5.02 to 44.27]

5. Secondary Outcome: Change From Baseline to Week 12 in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: The BASDAI is a validated self-reported instrument, which consists of six 10-unit horizontal Numeric Rating Scales (NRS) to measure severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration, respectively) over the last week. The final BASDAI score ranges from 0 to 10, with lower scores indicating lower disease activity.
  The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
  Note: Missing data was imputed using multiple imputation based on the Markov-Chain Monte Carlo method for the intermittent missing data, followed by monotone regression for the monotone missing data assuming missing at random.
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (FAS) | BKZ 16 mg (FAS) | BKZ 64 mg (FAS) | BKZ 160 mg (FAS) | BKZ 320 mg (FAS)
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 61
scores on a scale | -1.0 (0.38) | -1.6 (0.38) | -2.6 (0.38) | -2.6 (0.38) | -2.9 (0.38)
Statistical Analysis 1: Comparison: Placebo (FAS) vs BKZ 16 mg (FAS); [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.094, ANCOVA; LS Mean Difference vs placebo = -0.6, 95% CI 2-sided [-1.31 to 0.10], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: Placebo (FAS) vs BKZ 64 mg (FAS); [analysis description as in outcome 2, analysis 2]; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference vs placebo = -1.6, 95% CI 2-sided [-2.34 to -0.91], Standard Error of Mean 0.37
Statistical Analysis 3: Comparison: Placebo (FAS) vs BKZ 160 mg (FAS); [analysis description as in outcome 2, analysis 2]; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference vs placebo = -1.6, 95% CI 2-sided [-2.35 to -0.91], Standard Error of Mean 0.37
Statistical Analysis 4: Comparison: Placebo (FAS) vs BKZ 320 mg (FAS); [analysis description as in outcome 2, analysis 2]; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference vs placebo = -1.9, 95% CI 2-sided [-2.60 to -1.18], Standard Error of Mean 0.36

6. Secondary Outcome: Change From Baseline to Week 12 in the Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: The BASFI is a validated disease-specific instrument for assessing physical function. The BASFI comprises 10 items relating to the past week. The BASFI is the mean of the 10 scores such that the total score ranges from 0 (Easy) to 10 (Impossible), with lower scores indicating better physical function.
  The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
  Note: Missing data was imputed using multiple imputation based on the Markov-Chain Monte Carlo method for the intermittent missing data, followed by monotone regression for the monotone missing data assuming missing at random.
Time Frame: From Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (FAS) | BKZ 16 mg (FAS) | BKZ 64 mg (FAS) | BKZ 160 mg (FAS) | BKZ 320 mg (FAS)
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 61
scores on a scale | -0.7 (0.39) | -1.4 (0.38) | -1.8 (0.38) | -1.9 (0.38) | -2.2 (0.38)
Statistical Analysis 1: Comparison: Placebo (FAS) vs BKZ 16 mg (FAS); [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.075, ANCOVA; LS Mean Difference vs placebo = -0.6, 95% CI 2-sided [-1.35 to 0.07], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: Placebo (FAS) vs BKZ 64 mg (FAS); [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.003, ANCOVA; LS Mean Difference vs placebo = -1.1, 95% CI 2-sided [-1.79 to -0.37], Standard Error of Mean 0.36
Statistical Analysis 3: Comparison: Placebo (FAS) vs BKZ 160 mg (FAS); [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.002, ANCOVA; LS Mean Difference vs placebo = -1.1, 95% CI 2-sided [-1.84 to -0.42], Standard Error of Mean 0.36
Statistical Analysis 4: Comparison: Placebo (FAS) vs BKZ 320 mg (FAS); [analysis description as in outcome 2, analysis 2]; Test type: Other; p < 0.001, ANCOVA; LS Mean Difference vs placebo = -1.5, 95% CI 2-sided [-2.22 to -0.81], Standard Error of Mean 0.36

7. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE) During the Study
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From Screening until Safety Follow-Up Visit (up to Week 77)
Population: The SS consisted of all randomized participants who received at least 1 dose of IMP.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (SS) - up to Wk 12: This arm consisted of all participants who received placebo at any time in the study (up to Week 12). Participants formed the Safety Set (SS).
- BKZ 16 mg (SS) - up to Wk 12: This arm consisted of all participants who received bimekizumab (BKZ) 16 milligrams (mg) every 4 weeks (Q4W) at any time in the study (up to Week 12). Participants formed the SS.
- BKZ 64 mg (SS) - up to Wk 12: This arm consisted of all participants who received bimekizumab (BKZ) 64 mg every 4 weeks (Q4W) at any time in the study (up to Week 12). Participants formed the SS.
- BKZ 160 mg (SS) - up to Wk 73: This arm consisted of all participants who received bimekizumab (BKZ) 160 mg every 4 weeks (Q4W) at any time in the study (up to Week 73). Participants formed the SS.
- BKZ 320 mg (SS) - up to Wk 73: This arm consisted of all participants who received bimekizumab (BKZ) 320 mg every 4 weeks (Q4W) at any time in the study (up to Week 73). Participants formed the SS.
Arm/Group | Placebo (SS) - up to Wk 12 | BKZ 16 mg (SS) - up to Wk 12 | BKZ 64 mg (SS) - up to Wk 12 | BKZ 160 mg (SS) - up to Wk 73 | BKZ 320 mg (SS) - up to Wk 73
Number analyzed (Participants) | 60 | 61 | 58 | 149 | 150
percentage of participants | 45.0 | 44.3 | 34.5 | 69.8 | 82.0

8. Secondary Outcome: Percentage of Participants With at Least One Serious Adverse Event (SAE) During the Study
Description: A serious adverse event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalisation or prolongation of existing hospitalisation
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardise the patients, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Screening until Safety Follow-Up Visit (up to Week 77)
Population: The SS consisted of all randomized participants who received at least 1 dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) - up to Wk 12 | BKZ 16 mg (SS) - up to Wk 12 | BKZ 64 mg (SS) - up to Wk 12 | BKZ 160 mg (SS) - up to Wk 73 | BKZ 320 mg (SS) - up to Wk 73
Number analyzed (Participants) | 60 | 61 | 58 | 149 | 150
percentage of participants | 3.3 | 0 | 3.4 | 3.4 | 4.0

9. Secondary Outcome: Percentage of Participants Who Withdrew Due to an Adverse Event (AE) During the Study
Description: An AE is any untoward medical occurrence in a participant or trial subject that is administered a drug or biologic (medicinal product) or that is using a medical device.
  The event does not necessarily have a causal relationship with that treatment or usage. The results of this Secondary Outcome Measure were summarized from the adverse event pages of the Case Report Forms.
Time Frame: From Screening until Safety Follow-Up Visit (up to Week 77)
Population: The SS consisted of all randomized participants who received at least 1 dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) - up to Wk 12 | BKZ 16 mg (SS) - up to Wk 12 | BKZ 64 mg (SS) - up to Wk 12 | BKZ 160 mg (SS) - up to Wk 73 | BKZ 320 mg (SS) - up to Wk 73
Number analyzed (Participants) | 60 | 61 | 58 | 149 | 150
percentage of participants | 1.7 | 3.3 | 1.7 | 4.7 | 6.7

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from Baseline until the Safety Follow-Up Visit (up to Week 73)
Description: At Week 12, placebo, BKZ 16 mg and BKZ 64 mg subjects were re-randomized to either BKZ 160 mg or BKZ 320 mg. Subjects randomized to BKZ 160 mg group or BKZ 320 mg at Baseline were not re-randomized at Week 12 and remained on their original treatment. The Safety Set is based on actual treatment, other populations are based on planned treatment.
Arm/Group | Placebo (SS) - up to Wk 12 | BKZ 16 mg (SS) - up to Wk 12 | BKZ 64 mg (SS) - up to Wk 12 | BKZ 160 mg (SS) - up to Wk 73 | BKZ 320 mg (SS) - up to Wk 73
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/61 | 0/58 | 1/149 | 0/150
Serious Adverse Events (participants affected / at risk) | 2/60 | 0/61 | 2/58 | 5/149 | 6/150
Other Adverse Events (participants affected / at risk) | 2/60 | 2/61 | 4/58 | 42/149 | 56/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) - up to Wk 12 (N=60) | BKZ 16 mg (SS) - up to Wk 12 (N=61) | BKZ 64 mg (SS) - up to Wk 12 (N=58) | BKZ 160 mg (SS) - up to Wk 73 (N=149) | BKZ 320 mg (SS) - up to Wk 73 (N=150)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) - up to Wk 12 (N=60) | BKZ 16 mg (SS) - up to Wk 12 (N=61) | BKZ 64 mg (SS) - up to Wk 12 (N=58) | BKZ 160 mg (SS) - up to Wk 73 (N=149) | BKZ 320 mg (SS) - up to Wk 73 (N=150)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 8 (10) | 8 (11)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 6 (8)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 12 (12)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 13 (19) | 19 (22)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 5 (7) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT02963506/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT02963506/SAP_001.pdf